CLINICAL TRIAL: NCT06982859
Title: A Phase 1, Investigator- and Participant-Blinded Study to Evaluate the Effect of Retatrutide on α- and β- Cell Function and Insulin Sensitivity in Adult Participants With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Effect of Retatrutide on Insulin Secretion and Insulin Sensitivity in Adult Participants With Type 2 Diabetes Mellitus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27317; J1I-MC-GZQG (Other: Eli Lilly and Company); 2024-518470-13-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-14; First posted 2025-05-21 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus; Insulin Sensitivity
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — retatrutide; semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor is blinded to Retatrutide/Placebo. Semaglutide is open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Retatrutide (Experimental): Retatrutide administered subcutaneously (SC).
  Interventions: Drug: Retatrutide
- Semaglutide (Active Comparator): Semaglutide administered SC.
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Retatrutide — Administered SC
  Other Names: LY3437943
  Arms: Retatrutide
Drug: Semaglutide — Administered SC
  Arms: Semaglutide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The primary objective of Study GZQG is to compare the effect of retatrutide and placebo on total clamp disposition index (cDI) after 28 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with Type 2 Diabetes Mellitus (T2DM) for at least 6 months prior to screening.
* Treated with diet and exercise and metformin daily, with or without other allowed oral antihyperglycaemia medications (OAMs), 3 months prior to screening. Allowed OAMs are dipeptidyl peptidase-4 inhibitors (DPP-IV) inhibitors, sodium/glucose cotransporter 2 (SGLT2) inhibitors, glinides, and sulfonylureas.
* Have a HbA1c value at screening of:

  * 6.5% and ≤ 9.5 % if on metformin with or without SGLT2 inhibitors, or
  * 6% and ≤8.5% if on metformin in combination with allowed OAMs that require washout.
* Have venous access sufficient to allow for blood sampling as per the protocol.
* Have clinical laboratory test results within normal reference range for the population or investigative site or results with acceptable deviations that are judged to be not clinically significant by the investigator.
* Have a body mass index (BMI) between 25 kilograms per meter squared (kg/m²) and 45 kg/m², both inclusive, at screening.
* Have had a stable body weight that is less than 5% change during the 3-month period prior to screening.

Exclusion Criteria:

* Have Type 1 Diabetes Mellitus (T1DM)
* Have had more than 1 episode of severe hypoglycaemia, as defined by the American Diabetes Association criteria, within 6 months before screening or a history of hypoglycaemia unawareness or poor recognition of hypoglycaemic symptoms; any participant that cannot communicate an understanding of hypoglycaemic symptoms and the appropriate treatment of hypoglycaemia prior to the first dose of study drug should also be excluded.
* Have had 1 or more episodes of ketoacidosis or hyperosmolar state/coma requiring hospitalisation within the 6 months prior to screening.
* Are currently receiving, planning to receive, or in need of treatment, that is, intravitreal injections of Vascular Endothelial Growth Factor inhibitor or corticosteroids, focal/grid macular laser surgery, panretinal photocoagulation, or vitrectomy for diabetic retinopathy at screening.
* Have impaired renal estimated glomerular filtration rate <60.0 mL/min/1.73 m² calculated by Chronic Kidney Disease-Epidemiology (2021).
* Have acute or chronic pancreatitis or a history of acute idiopathic pancreatitis.
* Have elevations in:

  * serum aspartate aminotransferase (AST) >2.5X the upper limit of normal (ULN)
  * serum alanine aminotransferase (ALT) >2.5X ULN
  * total bilirubin level (TBL) >1.5X ULN (except, participants with Gilbert's syndrome), or
  * Alkaline phosphatase (ALP) level ≥1.5X ULN
* Show evidence of possible chronic or active hepatitis B, including hepatitis B core antibody and/or hepatitis B surface antigen positivity.
* Have a positive Hepatitis C virus (HCV) antibody (Ab) test. Participants with a positive HCV Ab test at screening can be included only if a confirmatory HCV ribonucleic acid (RNA) test is negative.
* Have a known clinically significant gastric emptying abnormality, have undergone gastric bypass (bariatric) surgery or restrictive bariatric surgery or chronically take drugs that directly affect GI motility.
* Have had within 3 months prior to screening:

  * acute myocardial infarction
  * congestive heart failure New York Heart Association (NYHA) class III or IV, and/or
  * cerebrovascular accident [stroke]
  * coronary artery revascularisation
  * hospitalization hospitalisation for unstable angina
  * hospitalization hospitalisation due to congestive heart failure.
* Have a history of additional risk factors for Torsades de Pointes (for example, heart failure, hypokalaemia, family history of Long QT Syndrome), as judged by the investigator.
* Have a 12-lead ECG abnormality at screening that, in the opinion of the investigator, increases the risks associated with participating in the study or may confound electrocardiogram (ECG) data analysis.
* Have a personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome Type 2 (MEN 2).
* Have an active or untreated malignancy or have been in remission from a clinically significant malignancy for <5 years prior to screening. Exceptions:

  * basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
  * cervical carcinoma in situ, with no evidence of recurrence within the 5 years prior to baseline, or
  * in situ prostate cancer.
* Have, in the opinion of the investigator, evidence of significant, uncontrolled endocrine abnormality, for example, thyrotoxicosis or adrenal crisis.
* Have a prior or planned surgical treatment for obesity.
* Have a prior or planned endoscopic and/or device-based therapy for obesity.
* Have taken any glucose-lowering medications other than metformin, DPP IV inhibitors, sulfonylureas and/or SGLT-2 inhibitors, regardless of the indication for use, any time within the 3 months prior to screening.
* Have taken prescribed or over-the-counter (OTC) medications, either approved or unapproved, or alternative remedies, including herbal or nutritional supplements, intended to promote body weight reduction, within 3 months prior to screening.
* Have evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies.
* Have a calcitonin level at screening of ≥35.0 nanograms per liter (ng/L), [≥35.0 picograms per milliliter (pg/mL)].

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Total Clamp Disposition Index (cDI) for Comparison of Retatrutide With Placebo | Baseline, Week 28
  Change from baseline in total cDI for comparison of retatrutide with placebo

SECONDARY OUTCOMES:
Change from Baseline in cDI for Comparison Between Retatrutide and Semaglutide | Baseline, Week 28
  Change from baseline in total cDI for comparison between retatrutide and semaglutide
Change from Baseline in Hyperinsulinemic Euglycemic Clamp M-value | Baseline, Week 28
  Change from baseline in hyperinsulinemic euglycemic clamp M-value
Change from Baseline in First Phase Incremental Insulin Secretion Rate (ISR) | Baseline, Week 28
  Change from baseline in first phase ISR.
Change from Baseline in Second Phase Total ISR | Baseline, Week 28
  Change from baseline in second phase total ISR
Change from Baseline in Total ISR | Baseline, Week 28
  Change from baseline in total ISR
Change from Baseline in Insulin Response to Arginine [Incremental Insulin Area Under the Curve (AUC) arginine, 0-10minutes] | Baseline, Week 28
  Change from baseline in insulin response to arginine [Incremental Insulin AUC arginine, 0-10minutes].
Change from Baseline in Insulin Response to Arginine (Incremental Insulin AUC arginine, 0-30minutes) | Baseline, Week 28
  Change from baseline in insulin response to arginine (Incremental Insulin AUC arginine, 0-30minutes).
Change from Baseline in Beta-cell (β-cell) Glucose Sensitivity (GS) | Baseline, Week 28
  Change from baseline in β-cell GS.
Change from Baseline in β-cell Glucose Sensitivity (GS) from Standardized Mixed-Meal Tolerance Test (sMMTT) | Baseline, Week 28
  Change from baseline in β-cell GS from sMMTT.
Change from Baseline in ISR at Fixed Glucose Concentration (ISRg) from sMMTT | Baseline, Week 28
  Change from baseline in ISR at fixed glucose concentration (ISRg) from sMMTT
Change from Baseline Fasting Glucose During sMMTT (Total and Incremental AUC0-240min) | Baseline, Week 28
  Change from baseline fasting glucose during sMMTT (total and incremental AUC0-240min)
Change from Baseline Postmeal Glucose During sMMTT (Total and Incremental AUC0-240min) | Baseline, Week 28
  Change from baseline postmeal glucose during sMMTT (total and incremental AUC0-240min)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Profil Institut für Stoffwechselforschung, Neuss, Germany

IPD SHARING:
Plan to Share IPD: No